CLINICAL TRIAL: NCT05679557
Title: Comprehensive Geriatric Assessment for Perioperative Optimization in Cystectomy
Acronym: COMPETENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); Aalborg University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jørgen Bjerggaard Jensen, Professor, DMSc, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-182-22
Record Dates: First submitted 2022-12-20; First posted 2023-01-11 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Bladder Cancer
Keywords: Frailty; Comprehensive Geriatric Assessment
MeSH Terms: conditions — Urinary Bladder Neoplasms; Frailty | interventions — Methods

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (No Intervention): Perioperative "care as usual" according to exciting principles and guidelines
- Geriatric (Experimental): Perioperative geriatric assessment and tailored interventions in relation to radical cystectomy.
  Interventions: Other: Perioperative geriatric assessment and intervention

INTERVENTIONS:
Other: Perioperative geriatric assessment and intervention — The intervention will comprise a preoperative, thorough geriatric, multidisciplinary assessment (CGA) and tailored interventions, focused on optimizing health issues of expected importance in further course of surgery. Furthermore, postoperative ward rounds by a geriatric team will be conducted. Thus, the course of treatment for each patient will be a close interdisciplinary collaboration.
  Arms: Geriatric

SUMMARY:
Patients with muscle-invasive bladder cancer are often older and multimorbid, thus in an increased risk of perioperative mortality and morbidity in relation to radical cystectomy (RC). The aim of the study is to investigate the effect of perioperative Comprehensive Geriatric Assessment (CGA) and tailored intervention in older, frail patients with bladder cancer undergoing RC.

DETAILED DESCRIPTION:
Patients will be randomized 1:1 and allocated into either control or intervention study arm. The control group will receive perioperative "care as usual" according to exciting principles and guidelines. The intervention will comprise a preoperative, thorough geriatric, multidisciplinary assessment, focused on optimizing health issues of expected importance in further course of surgery. Furthermore, postoperative ward rounds by a geriatric team will be conducted. Thus, the course of treatment for each patient will be a close interdisciplinary collaboration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with muscle-invasive bladder cancer and scheduled radical cystectomy.
2. Planned urinary diversion with an ileal conduit
3. Age ≥ 65 years.
4. Patients considered frail by G8 screening tool (total score ≤14).

Exclusion Criteria:

1. Patients who refuse or are not able to provide informed consent.
2. Patients who do not speak or understand Danish.
3. Planned concomitant nephroureterectomy or other major surgical intervention at the same time as RC

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Days Alive and out of Hospital (DAOH) | Within 90 days after cystectomy
  Primary outcome will be DAOH counted from day of surgery until 90 days after surgery. DAOH as an endpoint combines the duration of hospital stay, the burden of subsequently readmissions and mortality, and hence is an expression for the expected reduction in medical postoperative complications.

SECONDARY OUTCOMES:
Days Alive and out of Hospital (DAOH) | Within 30 days after cystectomy
  Secondary outcome will be DAOH counted from day of surgery until 30 days after surgery.
Complications | Within 30 and 90 days after cystectomy
  Number and severity (Clavien-Dindo grad I-V)
Length of stay | Within 90 days after surgery
  Number of days hospitalized during the index hospitalization
Hospital readmissions | Within 30 and 90 days after cystectomy
  Number of days admitted to hospital
Patient Quality of Life | Within 30 and 90 days postoperatively
  Quality of Life evaluated by the EuroQol 5D questionnaire (EQ-ED-5L)
Patient Quality of Life | Within 30 and 90 days postoperatively
  Quality of Life evaluated by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ C30/BLM30 (muscle invasive bladder cancer)).
Mortality | Within 30 and 90 days after cystectomy
  Number
Chair stand test (CST) | 3 weeks postoperatively
  Physical function measured by 30-s CST

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen S Bjerggaard Jensen, Prof., DMSc, Principal Investigator — Aarhus University Hospital and Aarhus University
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No